CLINICAL TRIAL: NCT02539550
Title: A Phase 1, Placebo-controlled, Randomized, Subject- And Investigator-blind, Sponsor-open, Crossover Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Pf-06266047 After Administration Of Single Ascending Doses To Healthy Adult Subjects
Brief Title: A Study To Evaluate the Safety, Tolerability, And Pharmacokinetics Of PF-06266047 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: B7481001; 2015-001796-52 (EudraCT Number)
Record Dates: First submitted 2015-08-10; First posted 2015-09-03 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: PF-06266047; safety; tolerability; pharmacokinetics; first-in-human; healthy volunteers; PDE4; phosphodiesterase-4

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-06266047 (Experimental): PF-06266047
  Interventions: Drug: PF-06266047

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PF-06266047 — PF-06266047
  Arms: PF-06266047

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of PF-06266047 after first-time administration to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non-childbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests. Female subjects of non-childbearing potential must meet at least one of the following criteria:

   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level confirming the post-menopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations) will be considered to be of childbearing potential.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Subject must be willing to avoid direct sunlight exposure or any high intensity ultraviolet light exposure, from the first day of dosing with study medication and until the follow-up visit; and to apply sun cream/lotion with a high sun protection factor, as appropriate.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug screen.
4. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
5. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer).
6. Screening supine blood pressure >140 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is >140 mm Hg (systolic) or >90 mm Hg (diastolic), the BP should be repeated two more times and the average of the three BP values should be used to determine the subject's eligibility.
7. Screening supine 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
8. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat, if deemed necessary:

   * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic aminotransferase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic aminotransferase (SGPT) >1.5 x upper limit of normal (ULN);
   * Total bilirubin >1.5 x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is <ULN.
9. Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product or longer based upon the compound's half-life characteristics.
10. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of <1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor. Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of study medication.
11. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
12. History of sensitivity to heparin or heparin-induced thrombocytopenia.
13. Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
14. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
15. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
16. Any subject considered at risk of suicide or self harm based on investigator judgement and/or the details of a risk assessment.
17. Use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Baseline up to 1 day of dosing
  Number of participants with AEs occurring after first dose of study drug. Relatedness to study drug will be assessed by investigator.
Number of subjects with standard safety laboratory test results of potential clinical significance | Baseline up to 1 day of dosing
  Number of subjects with standard safety laboratory test results of potential clinical significance (according to pre-defined criteria).
Electrocardiogram (ECG) | 0, 1, 2, 4, 8, 12, 24, 48, and 72 hours post-dose
  Absolute values and changes from baseline for the ECG parameters
Orthostatic blood pressure and pulse rate | 0, 1, 2, 4, 8, 12, 24, 48, and 72 hours post-dose
  Absolute values and changes from baseline for blood pressure and pulse rate
Abnormal rhythms as observed on continuous cardiac telemetry | Baseline period of at least 2 hours and continuous tracing for at least 8 hours following single dose administration
  All abnormal rhythms will be reviewed by the study physician for the presence of rhythms of potential clinical concern. The time, duration and description of any clinically significant event will be recorded.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  Maximum Observed Plasma Concentration (Cmax)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0, 0.5, 1.5, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, and 72 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7481001&StudyName=A%20Phase%201%2C%20Placebo-controlled%2C%20Randomized%2C%20Subject-%20And%20Investigator-blind%2C%20Sponsor-open%2C%20Crossover%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetics%20Of%20Pf-06266047%20After%20Administration%20Of%20Single%20Ascending%20Doses%20To%20Healthy%20Adult%20Subjects